CLINICAL TRIAL: NCT02410161
Title: Effect of an Alpha-linolenic Acid-rich Supplement on Ketogenesis and Plasma n-3 Polyunsaturated Fatty Acids in Young Compared to Older Adults
Brief Title: Effect of an Alpha-linolenic Acid-rich Supplement on Ketogenesis and Plasma Fatty Acids
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2014-389
Record Dates: First submitted 2015-03-16; First posted 2015-04-07 (Estimated); Results first posted 2019-02-18 (Actual); Last update posted 2019-02-18 (Actual); Status verified 2015-03

CONDITIONS: Healthy
Keywords: ketone; α-linolenic acid; flaxseed; aging; β-hydroxybutyrate; acetoacetate; omega-3 fatty acids; ketogenesis
MeSH Terms: conditions — Ketosis

STUDY DESIGN:
Intervention Model Description: Dietary Supplement: alpha-linolenic acid-rich supplement
Oversight: Data Monitoring Committee: No

ARMS (1):
- 4 week ALA treatment (Experimental): Participants will receive the alpha-linolenic acid-rich supplement (1000mg 4 times par day) for 4 weeks
  Interventions: Dietary Supplement: alpha-linolenic acid-rich supplement

INTERVENTIONS:
Dietary Supplement: alpha-linolenic acid-rich supplement — each participant consumed one 1000 mg capsule of flaxseed oil four times per day for 4 weeks, providing a total of 2 g/d of ALA. The capsules used were a commercially available flaxseed oil supplement containing ALA at 56% of total fatty acids (Jamieson, Toronto, ON, Canada). The other main fatty acids present in flaxseed oil include linoleic acid (18%), oleic acid (16%), palmitic and stearic acid (10% combined).

SUMMARY:
Background: As the main alternative fuel to glucose for the brain, increased plasma ketones could potentially help compensate for brain glucose hypometabolism occurring during aging. The precursor long-chain n-3 polyunsaturated fatty acid (PUFA), α-linolenic acid (ALA), is normally mostly β-oxidized and so could potentially be used to stimulate ketogenesis in humans.

Objective: To compare the impact of an ALA-rich supplement on the ketogenic response in young and older healthy adults.

Design: Ten young and ten older adults will consume a flaxseed oil supplement providing 2 g/d of ALA for 4 weeks. Plasma ketones, free fatty acids, triglycerides, glucose and insulin will be measured over 6 h during two metabolic study days, one before and one at the end of the supplementation.

Hypothesis: ALA-rich supplement for 4 weeks will increase ketone production in both groups.

ELIGIBILITY:
Inclusion Criteria:

* aged between 18 and 30 or 65 years and more

Exclusion Criteria:

* non smoker
* pregnancy or breastfeeding
* diabetes or insulin resistance
* uncontrolled thyroid disease, hepatic or renal disease
* uncontrolled high blood pressure
* medical treatment influencing lipid or glucide metabolism
* ongoing or past severe drug or alcohol abuse
* dementia or psychiatric difficulties or depression
* chronic immune condition or inflammation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-07; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Cunnane, PhD, Principal Investigator — Université de Sherbrooke

RESULTS

PARTICIPANT FLOW:
Groups:
- Young Group 4 Week ALA Treatment: Participants will receive the alpha-linolenic acid-rich supplement (ALA) (1000mg 4 times par day) for 4 weeks
  alpha-linolenic acid-rich supplement: each participant consumed one 1000 mg capsule of flaxseed oil four times per day for 4 weeks, providing a total of 2 g/d of ALA. The capsules used were a commercially available flaxseed oil supplement containing ALA at 56% of total fatty acids (Jamieson, Toronto, ON, Canada). The other main fatty acids present in flaxseed oil include linoleic acid (18%), oleic acid (16%), palmitic and stearic acid (10% combined).
- Old Group 4 Week ALA Treatment: Participants will receive the alpha-linolenic acid-rich supplement (1000mg 4 times par day) for 4 weeks
  alpha-linolenic acid-rich supplement: each participant consumed one 1000 mg capsule of flaxseed oil four times per day for 4 weeks, providing a total of 2 g/d of ALA. The capsules used were a commercially available flaxseed oil supplement containing ALA at 56% of total fatty acids (Jamieson, Toronto, ON, Canada). The other main fatty acids present in flaxseed oil include linoleic acid (18%), oleic acid (16%), palmitic and stearic acid (10% combined).
Period: Overall Study
Arm/Group | Young Group 4 Week ALA Treatment | Old Group 4 Week ALA Treatment
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Young Group 4 Week ALA Treatment; Old Group 4 Week ALA Treatment: Participants will receive the alpha-linolenic acid-rich supplement (1000mg 4 times par day) for 4 weeks
  alpha-linolenic acid-rich supplement: each participant consumed one 1000 mg capsule of flaxseed oil four times per day for 4 weeks, providing a total of 2 g/d of ALA. The capsules used were a commercially available flaxseed oil supplement containing ALA at 56% of total fatty acids (Jamieson, Toronto, ON, Canada). The other main fatty acids present in flaxseed oil include linoleic acid (18%), oleic acid (16%), palmitic and stearic acid (10% combined).
- Total: Total of all reporting groups
Arm/Group | Young Group 4 Week ALA Treatment | Old Group 4 Week ALA Treatment | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 0 | 10
  >=65 years | 0 | 10 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 25 (2.8) | 73 (7) | 52 (25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 13
  Male | 4 | 3 | 7
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Ketone Production
Description: Total Ketone (acetoacetate + beta-hydroxybutyrate) concentration in plasma in average during the metabolic study day, measured hourly between 1 and 6h after breakfast
Time Frame: After 4 weeks
Measure: Mean (Standard Error); unit: µmol/L
Arm/Group | Young Group 4 Week ALA Treatment | Old Group 4 Week ALA Treatment
Number analyzed (Participants) | 10 | 10
µmol/L | 217.71 (24) | 187.48 (17)

2. Secondary Outcome: Plasma Glucose
Description: Glucose measured in plasma in average during the metabolic study day, measure hourly between 0 and 6 h after breakfast
Time Frame: After 4 weeks
Measure: Mean (Standard Error); unit: mmol/L
Arm/Group | Young Group 4 Week ALA Treatment | Old Group 4 Week ALA Treatment
Number analyzed (Participants) | 10 | 10
mmol/L | 4.75 (0.13) | 5.46 (0.19)

3. Secondary Outcome: Plasma Triglycerides
Description: Triglycerides measured in plasma in average during the metabolic study day, measured hourly between 1 to 6h after breakfast
Time Frame: After 4 weeks
Measure: Mean (Standard Error); unit: mmol/L
Arm/Group | Young Group 4 Week ALA Treatment | Old Group 4 Week ALA Treatment
Number analyzed (Participants) | 10 | 10
mmol/L | 0.97 (0.15) | 1.81 (0.29)

4. Secondary Outcome: Plasma Free Fatty Acids
Description: Free fatty acids measured in plasma in average during the metabolic study day, measured hourly between 1 to 6h after breakfast
Time Frame: 4 weeks
Measure: Mean (Standard Error); unit: mmol/L
Arm/Group | Young Group 4 Week ALA Treatment | Old Group 4 Week ALA Treatment
Number analyzed (Participants) | 10 | 10
mmol/L | 0.48 (0.05) | 0.55 (0.04)

5. Secondary Outcome: Insulin Concentration in Plasma
Description: Insulin measured in plasma in average during the metabolic study day, measured hourly between 0 ans 6 h after breakfast
Time Frame: after 4 weeks
Measure: Mean (Standard Error); unit: µIU/mL
Arm/Group | Young Group 4 Week ALA Treatment | Old Group 4 Week ALA Treatment
Number analyzed (Participants) | 10 | 10
µIU/mL | 10.48 (1.48) | 14.87 (2.63)

ADVERSE EVENTS:
Time Frame: Adverse event were collected during the 4-weeks supplementation of each participant
Arm/Group | Young Group 4 Week ALA Treatment | Old Group 4 Week ALA Treatment
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes